CLINICAL TRIAL: NCT02482571
Title: Metabolic Changes in the Activated Human Visual Cortex During Mild Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201503M65382
Record Dates: First submitted 2015-06-23; First posted 2015-06-26 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Brain Hypoxia
Keywords: Functional MRS; Glutamate
MeSH Terms: conditions — Hypoxia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mild Hypoxia (Experimental): Subjects are exposed to an intervention that controls the composition of breathed air by using a gas blender (RespirAct). Subjects undergo MRI and MRS while breathing air with both normal oxygen concentration (normoxia) and reduced oxygen concentration (mild hypoxia).
  Interventions: Device: Mild Hypoxia

INTERVENTIONS:
Device: Mild Hypoxia — During normoxia, the computer-controlled gas blender provides a gas mixture that generates pressures of expired O2 and CO2 similar to the resting values measured for each subject (32-35mmHg and 100-110 mmHg, respectively). During mild hypoxia, we will target the same expired CO2 of normoxia and a 60 mmHg reduction of expired O2 from the resting value (to a minimum limit of 50 mmHg), which is expected to reduce arterial oxygen saturation to 82-85%. In mild hypoxia, the fraction of inspired oxygen is reduced from ~21% (room air) to ~12% (equivalent to an altitude of 4000 meters). During both conditions of normoxia and mild hypoxia, the brain activity of subjects is monitored with functional magnetic resonance spectroscopy (fMRS) while they are presented with visual stimuli.

SUMMARY:
The primary objective of this research is to measure changes in neurochemical concentrations during stimulation of the primary visual cortex, in both conditions of normoxia (normal oxygen availability) and induced mild hypoxia (reduced oxygen availability).

DETAILED DESCRIPTION:
The goal is to determine the effect of mild hypoxia on human brain energy metabolism of healthy young adult subjects. For this purpose, the Investigator will utilize non-invasive imaging modalities based on functional magnetic resonance spectroscopy (fMRS) to estimate metabolic changes during a visual stimulus, while subjects are exposed to well-controlled gas mixtures that resembles conditions of either normoxia or mild hypoxia. Identifying the impact of mild hypoxia on functional brain energy metabolism in the healthy human brain is a crucial step for generating hypotheses in multiple patient populations that experience mild hypoxia as consequence of their pathological condition, such as in sleep apnea and traumatic brain injury. The Investigator hypothesize that the energetic demands of neuronal activation as revealed by fMRS will not be affected by mild hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Those volunteers who are evaluated as normal and not met exclusion criteria will be potential candidates for this study.

Exclusion Criteria:

* Subjects with any type of bio-implant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc.).
* Subjects with any type of ferromagnetic bio-implant that could potentially be displaced or damaged, such as aneurysm clips, metallic skull plates, etc.
* Females.
* Subjects that exhibit noticeable anxiety and/or claustrophobia.
* Subjects who cannot adhere to the experimental protocol for any reason.
* Subjects who have cardiac or known circulatory impairment, and/or the inability to perspire (poor thermoregulatory function).
* Subjects who have known conditions which can lead to emergency medical care.
* Been diagnosed by a physician as having a psychiatric disorder, substance abuse, neurological, cardiovascular.
* Been diagnosed by a physician as having respiratory diseases.
* Had a brain tumor or stroke.
* Started taking chemotherapy or immunomodulatory agents, or had any radiation treatment that could affect the brain.
* Had two or more seizures, or been given a diagnosis of epilepsy.
* Gotten a non-removable piercing or permanent eyeliner.
* Had a head injury that caused you to lose consciousness for more than 30 minutes or have amnesia for more than 24 hours.
* Anyone with a history of sleep apnea or head trauma that may have caused Traumatic Brain Injury (TBI).
* Gotten some type of metal in your body, either from a medical procedure or an injury.
* Male subjects with long beard which wouldn't allow a complete seal between the mask and the face.
* Anyone who is not able to see long distance without glasses or contacts.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Mangia, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Center for Magnetic Resoance Research, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho YC, Vidyasagar R, Shen Y, Balanos GM, Golay X, Kauppinen RA. The BOLD response and vascular reactivity during visual stimulation in the presence of hypoxic hypoxia. Neuroimage. 2008 Jun;41(2):179-88. doi: 10.1016/j.neuroimage.2008.02.048. Epub 2008 Mar 6. PMID 18396415
- [Background] Tuunanen PI, Murray IJ, Parry NR, Kauppinen RA. Heterogeneous oxygen extraction in the visual cortex during activation in mild hypoxic hypoxia revealed by quantitative functional magnetic resonance imaging. J Cereb Blood Flow Metab. 2006 Feb;26(2):263-73. doi: 10.1038/sj.jcbfm.9600186. PMID 16079793
- See also: Profile of Principle Investigator — http://www.cmrr.umn.edu/facultystaff/mangia.shtml

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Hypoxia: Mild Hypoxia: During normoxia, the computer-controlled gas blender provides a gas mixture that generates pressures of expired O2 and CO2 similar to the resting values measured for each subject (32-35mmHg and 100-110 mmHg, respectively). During mild hypoxia, we will target the same expired CO2 of normoxia and a 60 mmHg reduction of expired O2 from the resting value (to a minimum limit of 50 mmHg), which is expected to reduce arterial oxygen saturation to 82-85%. In mild hypoxia, the fraction of inspired oxygen is reduced from ~21% (room air) to ~12%. During both conditions of normoxia and mild hypoxia, the brain activity of subjects is monitored with functional MRI (fMRI) and functional MRS (fMRS) during visual stimuli.
Period: Overall Study
Arm/Group | Mild Hypoxia
Started | 25
Completed | 17
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Scanner or Respiract failure | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Mild Hypoxia
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Glutamate Concentration During a Visual Stimulus Measured by fMRS at Normoxia
Description: Relative change in glutamate concentration from rest to visual stimulation as measured by fMRS (with water suppression) in the primary visual cortex during conditions of normoxia.
Time Frame: Baseline and Visual Stimulation at 4 minutes
Population: Out of the 17 experimental sessions that were successfully completed, 4 had data of insufficient quality. Therefore, a total of 13 sessions was used for final analyses.
Measure: Mean (Standard Deviation); unit: percentage of concentration (micromol/g)
Arm/Group | Mild Hypoxia
Number analyzed (Participants) | 13
percentage of concentration (micromol/g) | 4 (2.4)

2. Primary Outcome: Change in Glutamate Concentration During a Visual Stimulus Measured by Functional MRS at Hypoxia
Description: Relative change in glutamate concentration from rest to visual stimulation as measured by fMRS (with water suppression) in the primary visual cortex during conditions of hypoxia.
Time Frame: Baseline and Visual Stimulation at 4 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of concentration (micromol/g)
Arm/Group | Mild Hypoxia
Number analyzed (Participants) | 13
percentage of concentration (micromol/g) | 2.9 (1.9)

3. Secondary Outcome: Brain Activity Measured by Blood Oxygenation Level Dependent (BOLD) Signal at Normoxia
Description: Relative change in water signal intensity from rest to visual stimulation as measured by fMRS (without water suppression) in the primary visual cortex during conditions of normoxia.
Time Frame: Baseline and Visual Stimulation at 30 seconds
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal intensity
Groups:
- Mild Hypoxia: Mild Hypoxia: During normoxia, the computer-controlled gas blender provides a gas mixture that generates pressures of expired O2 and CO2 similar to the resting values measured for each subject (32-35mmHg and 100-110 mmHg, respectively). During mild hypoxia, we will target the same expired CO2 of normoxia and a 60 mmHg reduction of expired O2 from the resting value (to a minimum limit of 50 mmHg), which is expected to reduce arterial oxygen saturation to 82-85%. In mild hypoxia, the fraction of inspired oxygen is reduced from ~21% (room air) to ~12% . During both conditions of normoxia and mild hypoxia, the brain activity of subjects is monitored with functional MRI (fMRI) and functional MRS (fMRS) during visual stimuli.
Arm/Group | Mild Hypoxia
Number analyzed (Participants) | 13
percentage of signal intensity | 3.3 (2.0)

4. Secondary Outcome: Brain Activity Measured by Blood Oxygenation Level Dependent (BOLD) Signal at Hypoxia
Description: Relative change in water signal intensity from rest to visual stimulation as measured by fMRS (without water suppression) in the primary visual cortex during conditions of hypoxia.
Time Frame: Baseline and Visual Stimulation at 30 seconds
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of signal intensity
Arm/Group | Mild Hypoxia
Number analyzed (Participants) | 13
percentage of signal intensity | 1.2 (1.2)

ADVERSE EVENTS:
Groups:
- Mild Hypoxia: Mild Hypoxia: During normoxia, the computer-controlled gas blender provides a gas mixture that generates pressures of expired O2 and CO2 similar to the resting values measured for each subject (32-35mmHg and 100-110 mmHg, respectively). During mild hypoxia, we will target the same expired CO2 of normoxia and a 60 mmHg reduction of expired O2 from the resting value (to a minimum limit of 50 mmHg), which is expected to reduce arterial oxygen saturation to 82-85%. In mild hypoxia, the fraction of inspired oxygen is reduced from ~21% (room air) to ~12% (equivalent to an altitude of 4000 meters). During both conditions of normoxia and mild hypoxia, the brain activity of subjects is monitored with functional MRI (fMRI) and functional MRS (fMRS) during visual stimuli.
Arm/Group | Mild Hypoxia
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hypoxia (N=25)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle cramps in hands and tongue numbness
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mild Hypoxia (N=25)
Claustropobia (Psychiatric disorders) | 2 — Feeling of claustrophobia inside the MRI scanner
Nervousness (Psychiatric disorders) | 8 — Feeling nervous inside the MRI scanner and/or breathing through the mask
Sleepiness (General disorders) | 6 — Feeling sleepy inside the restricted and dark environment of the MRI scanner
Lightheadedness (General disorders) | 2 — Some lightheadedness while breathing through the mask at specific breathing pattern, or while just being inside the MRI scanner
Metallic Taste (General disorders) | 2 — Metallic taste inside the MRI scanner
Cold (General disorders) | 4 — Feeling cold inside the MRI scanner
Warmth (General disorders) | 2 — Feeling warm inside the MRI scanner

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No